CLINICAL TRIAL: NCT02456740
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of AMG 334 in Migraine Prevention
Brief Title: Study to Evaluate the Efficacy and Safety of Erenumab (AMG 334) in Migraine Prevention
Acronym: STRIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120296; 2014-004464-38 (EudraCT Number)
Record Dates: First submitted 2015-05-14; First posted 2015-05-28 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Migraine
Keywords: Migraine; Headache; Prevention; Prophylaxis
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo once a month (QM) by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase. At week 24, participants were re-randomized to receive either erenumab 70 mg or erenumab 140 mg, administered QM at weeks 24, 28, 32, 36, 40, 44, and 48, with actual dose blinded.
  Interventions: Drug: Placebo
- Erenumab 70 mg QM (Experimental): Participants received erenumab 70 mg QM by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase. At week 24, participants were re-randomized to receive either erenumab 70 mg or erenumab 140 mg, administered QM at weeks 24, 28, 32, 36, 40, 44, and 48, with actual dose blinded.
  Interventions: Drug: Erenumab
- Erenumab 140 mg QM (Experimental): Participants received erenumab 140 mg QM by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase. At week 24, participants were re-randomized to receive either erenumab 70 mg or erenumab 140 mg, administered QM at weeks 24, 28, 32, 36, 40, 44, and 48, with actual dose blinded.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Administered by subcutaneous injection once a month
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab 140 mg QM; Erenumab 70 mg QM
Drug: Placebo — Administered by subcutaneous injection once a month
  Arms: Placebo

SUMMARY:
The primary objective of the study was to evaluate the effect of erenumab compared to placebo on the change from baseline in monthly migraine days.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. The trial consisted of four phases: screening (≤ 3 weeks of initial screening and a 4-week baseline phase); the double-blind treatment phase (24 weeks) in which participants received placebo or erenumab 70 mg or 140 mg daily; the active-treatment phase, in which participants underwent repeat randomization and were assigned to receive 70 mg or 140 mg of erenumab (28 weeks); and a safety follow-up phase (12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* History of migraine (with or without aura) for ≥ 12 months prior to screening according to the International Headache Society (IHS) International Classification of Headache Disorders (ICHD-3) classification
* Migraine frequency: ≥ 4 and < 15 migraine days per month on average across the 3 months prior to screening and during baseline
* Headache frequency: < 15 headache days per month on average across the 3 months prior to screening and baseline
* Demonstrated at least 80% compliance with the eDiary.

Exclusion Criteria:

* Older than 50 years of age at migraine onset
* History of cluster headache or hemiplegic migraine headache
* Unable to differentiate migraine from other headache
* No therapeutic response with > 2 medication categories for prophylactic treatment of migraine after an adequate therapeutic trial
* Used a prohibited medication, device, or procedure within 2 months prior to the start of the baseline phase or during the baseline phase
* Concomitant use of 2 or more medications with possible migraine prophylactic effects within 2 months prior to the start of the baseline phase or during the baseline phase. If only 1 prophylactic medication is used, the dose must be stable within 2 months prior to the start of the baseline phase and throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (119):
- United States (58):
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Encino, California
  - Research Site, Irvine, California
  - Research Site, Los Alamitos, California
  - Research Site, Newport Beach, California
  - Research Site, Rancho Mirage, California
  - Research Site, Redlands, California
  - Research Site, Sherman Oaks, California
  - Research Site, Simi Valley, California
  - Research Site, Spring Valley, California
  - Research Site, Boulder, Colorado
  - Research Site, East Hartford, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sunrise, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Evansville, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Edgewood, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, New Bedford, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Plymouth, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Amherst, New York
  - Research Site, Plainview, New York
  - Research Site, Rochester, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Willoughby Hills, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Cumberland, Rhode Island
  - Research Site, Port Royal, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, West Jordan, Utah
  - Research Site, Charlottesville, Virginia
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Liège
  - Research Site, Lodelinsart
- Canada (5):
  - Research Site, Surrey, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Lévis, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Pardubice
  - Research Site, Prague
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Turku
- Germany (12):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hellersdorf
  - Research Site, Hüttenberg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Wiesbaden
  - Research Site, Würzburg
- Research Site, Leiden, Netherlands
- Poland (6):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Świdnik
  - Research Site, Warsaw
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Komárno
  - Research Site, Lučenec
- Sweden (4):
  - Research Site, Falköping
  - Research Site, Helsingborg
  - Research Site, Stockholm
  - Research Site, Uddevalla
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (7):
  - Research Site, Glasgow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Northwood
  - Research Site, Oxford
  - Research Site, Sidcup
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Background] Buse DC, Lipton RB, Hallstrom Y, Reuter U, Tepper SJ, Zhang F, Sapra S, Picard H, Mikol DD, Lenz RA. Migraine-related disability, impact, and health-related quality of life among patients with episodic migraine receiving preventive treatment with erenumab. Cephalalgia. 2018 Sep;38(10):1622-1631. doi: 10.1177/0333102418789072. Epub 2018 Aug 7. PMID 30086681
- [Background] Cheng S, Picard H, Zhang F, Eisele O, Mikol DD. Efficacy and safety of erenumab for migraine prevention: an overview. Japanese Journal of Headache. 2019; 45 : 493-505.
- [Background] Goadsby PJ, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Zhang F, Sapra S, Picard H, Mikol DD, Lenz RA. A Controlled Trial of Erenumab for Episodic Migraine. N Engl J Med. 2017 Nov 30;377(22):2123-2132. doi: 10.1056/NEJMoa1705848. PMID 29171821
- [Background] Zhou Y, Zhang F, Starcevic Manning M, Hu Z, Hsu CP, Chen PW, Peng C, Loop B, Mytych DT, Paiva da Silva Lima G. Immunogenicity of erenumab: A pooled analysis of six placebo-controlled trials with long-term extensions. Cephalalgia. 2022 Jul;42(8):749-760. doi: 10.1177/03331024221075621. Epub 2022 Mar 10. PMID 35272533
- [Background] Kawata AK, Ladd MK, Lipton RB, Buse DC, Bensink M, Shah S, Hareendran A, Mannix S, Mikol D. Reducing the physical, social, and emotional impact of episodic migraine: Results from erenumab STRIVE and ARISE phase III randomized trials. Headache. 2022 Feb;62(2):159-168. doi: 10.1111/head.14258. Epub 2022 Feb 8. PMID 35137394
- [Background] McAllister PJ, Turner I, Reuter U, Wang A, Scanlon J, Klatt J, Chou DE, Paiva da Silva Lima G. Timing and durability of response to erenumab in patients with episodic migraine. Headache. 2021 Nov;61(10):1553-1561. doi: 10.1111/head.14233. Epub 2021 Nov 28. PMID 34841526
- [Background] Ashina M, Kudrow D, Reuter U, Dolezil D, Silberstein S, Tepper SJ, Xue F, Picard H, Zhang F, Wang A, Zhou Y, Hong F, Klatt J, Mikol DD. Long-term tolerability and nonvascular safety of erenumab, a novel calcitonin gene-related peptide receptor antagonist for prevention of migraine: A pooled analysis of four placebo-controlled trials with long-term extensions. Cephalalgia. 2019 Dec;39(14):1798-1808. doi: 10.1177/0333102419888222. Epub 2019 Nov 10. PMID 31707815
- [Background] Kudrow D, Pascual J, Winner PK, Dodick DW, Tepper SJ, Reuter U, Hong F, Klatt J, Zhang F, Cheng S, Picard H, Eisele O, Wang J, Latham JN, Mikol DD. Vascular safety of erenumab for migraine prevention. Neurology. 2020 Feb 4;94(5):e497-e510. doi: 10.1212/WNL.0000000000008743. Epub 2019 Dec 18. PMID 31852816
- [Background] Lipton RB, Dodick DW, Kudrow D, Reuter U, Tenenbaum N, Zhang F, Lima GPDS, Chou DE, Mikol DD. Reduction in migraine pain intensity in patients treated with erenumab: A post hoc analysis of two pivotal randomized studies. Cephalalgia. 2021 Dec;41(14):1458-1466. doi: 10.1177/03331024211028966. Epub 2021 Aug 18. PMID 34407654
- [Background] Yucel A, Thach A, Kumar S, Loden C, Bensink M, Goldfarb N. Estimating the economic burden of migraine on US employers. Am J Manag Care. 2020 Dec 1;26(12):e403-e408. doi: 10.37765/ajmc.2020.88547. PMID 33315334
- [Derived] Lampl C, Kraus V, Lehner K, Loop B, Chehrenama M, Maczynska Z, Ritter S, Klatt J, Snellman J. Safety and tolerability of erenumab in individuals with episodic or chronic migraine across age groups: a pooled analysis of placebo-controlled trials. J Headache Pain. 2022 Aug 18;23(1):104. doi: 10.1186/s10194-022-01470-4. PMID 35978286
- [Derived] Ashina M, Goadsby PJ, Dodick DW, Tepper SJ, Xue F, Zhang F, Brennan F, Paiva da Silva Lima G. Assessment of Erenumab Safety and Efficacy in Patients With Migraine With and Without Aura: A Secondary Analysis of Randomized Clinical Trials. JAMA Neurol. 2022 Feb 1;79(2):159-168. doi: 10.1001/jamaneurol.2021.4678. PMID 34928306
- [Derived] Tepper SJ, Ashina M, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Picard H, Cheng S, Chou DE, Zhang F, Klatt J, Mikol DD. Reduction in acute migraine-specific and non-specific medication use in patients treated with erenumab: post-hoc analyses of episodic and chronic migraine clinical trials. J Headache Pain. 2021 Jul 23;22(1):81. doi: 10.1186/s10194-021-01292-w. PMID 34301173
- [Derived] Diener HC, Ashina M, Ritter S, Paiva Da Silva Lima G, Rasmussen S, Zielman R, Tfelt-Hansen P. Erenumab prevents the occurrence of migraine attacks and not just migraine days: Post-hoc analyses of a phase III study. Cephalalgia. 2021 Oct;41(11-12):1262-1267. doi: 10.1177/03331024211010308. Epub 2021 May 3. PMID 33939497
- [Derived] Broessner G, Reuter U, Bonner JH, Dodick DW, Hallstrom Y, Picard H, Zhang F, Lenz RA, Klatt J, Mikol DD. The Spectrum of Response to Erenumab in Patients With Episodic Migraine and Subgroup Analysis of Patients Achieving >/=50%, >/=75%, and 100% Response. Headache. 2020 Oct;60(9):2026-2040. doi: 10.1111/head.13929. Epub 2020 Aug 26. PMID 32851644
- [Derived] Pavlovic JM, Paemeleire K, Gobel H, Bonner J, Rapoport A, Kagan R, Zhang F, Picard H, Mikol DD. Efficacy and safety of erenumab in women with a history of menstrual migraine. J Headache Pain. 2020 Aug 3;21(1):95. doi: 10.1186/s10194-020-01167-6. PMID 32746775
- [Derived] Goadsby PJ, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Zhang F, Wright IK, Chou DE, Klatt J, Picard H, Lenz RA, Mikol DD. One-year sustained efficacy of erenumab in episodic migraine: Results of the STRIVE study. Neurology. 2020 Aug 4;95(5):e469-e479. doi: 10.1212/WNL.0000000000010019. Epub 2020 Jul 7. PMID 32636324
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 121 centers in Canada, Austria, Belgium, Czech Republic, Finland, Germany, Poland, Slovakia, Sweden, the United Kingdom, Turkey, the Netherlands and USA.
  The study consisted of a 24-week double-blind treatment phase and a 28-week active treatment phase.
Pre-assignment Details: At the end of the baseline phase, participants were randomized 1:1:1 to receive placebo, erenumab 70 mg, or erenumab 140 mg monthly for 24 weeks. Randomization was stratified by region and treatment status with migraine prophylactic medication.
  Participants were re-randomized at week 24 to erenumab 70 mg or 140 mg for 28 weeks.
Groups:
- Placebo: Participants received placebo once a month (QM) by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase.
- Erenumab 70 mg QM: Participants received erenumab 70 mg QM by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase.
- Erenumab 140 mg QM: Participants received erenumab 140 mg QM by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase.
- Placebo / Erenumab 70 mg: Participants originally randomized to receive placebo in the 24-week double-blind treatment phase were re-randomized at week 24 to receive erenumab 70 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
- Erenumab 70 mg / Erenumab 70 mg: Participants originally randomized to receive erenumab 70 mg QM in the 24-week double-blind treatment phase were re-randomized at week 24 to receive erenumab 70 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
- Erenumab 140 mg / Erenumab 70 mg: Participants originally randomized to receive erenumab 140 mg QM in the 24-week double-blind treatment phase were re-randomized at week 24 to receive erenumab 70 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
- Placebo / Erenumab 140 mg: Participants originally randomized to receive placebo QM in the 24-week double-blind treatment phase were re-randomized at week 24 to receive erenumab 140 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
- Erenumab 70 mg / Erenumab 140 mg: Participants originally randomized to receive erenumab 70 mg QM in the 24-week double-blind treatment phase were re-randomized at week 24 to receive erenumab 140 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
- Erenumab 140 mg / Erenumab 140 mg: Participants originally randomized to receive erenumab 140 mg QM in the 24-week double-blind treatment phase were re-randomized at week 24 to receive erenumab 140 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
Period: Double-blind Treatment Phase (24 Weeks)
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM | Placebo / Erenumab 70 mg | Erenumab 70 mg / Erenumab 70 mg | Erenumab 140 mg / Erenumab 70 mg | Placebo / Erenumab 140 mg | Erenumab 70 mg / Erenumab 140 mg | Erenumab 140 mg / Erenumab 140 mg
Started | 319 | 317 | 319 | 0 | 0 | 0 | 0 | 0 | 0
Received Study Drug | 319 | 314 | 319 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 282 | 284 | 292 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 37 | 33 | 27 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Decision by Sponsor | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 27 | 28 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Phase (Weeks 24 - 52)
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM | Placebo / Erenumab 70 mg | Erenumab 70 mg / Erenumab 70 mg | Erenumab 140 mg / Erenumab 70 mg | Placebo / Erenumab 140 mg | Erenumab 70 mg / Erenumab 140 mg | Erenumab 140 mg / Erenumab 140 mg
Started (Fourteen participants who completed the DBTP did not continue onto the active treatment phase) | 0 | 0 | 0 | 138 | 140 | 143 | 140 | 140 | 144
Completed | 0 | 0 | 0 | 124 | 123 | 130 | 131 | 128 | 126
Not Completed | 0 | 0 | 0 | 14 | 17 | 13 | 9 | 12 | 18
Not completed — Protocol Specified Criteria | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 10 | 11 | 9 | 8 | 8 | 9
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 2 | 4 | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM | Total
Number analyzed (Participants) | 319 | 317 | 319 | 955
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.2) | 41.1 (11.3) | 40.4 (11.1) | 40.9 (11.2)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 317 | 317 | 317 | 951
  65 - 74 years | 2 | 0 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 268 | 272 | 814
  Male | 45 | 49 | 47 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 26 | 22 | 80
  Not Hispanic or Latino | 287 | 291 | 297 | 875
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 8 | 5 | 4 | 17
  Black or African American | 24 | 24 | 18 | 66
  Multiple | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  White | 277 | 281 | 293 | 851
  Other | 6 | 6 | 2 | 14
Region [Count of Participants; unit: Participants]
  North America | 158 | 159 | 160 | 477
  Other | 161 | 158 | 159 | 478
Treatment Status with Migraine Prophylactic Medication [Count of Participants; unit: Participants]
  Current migraine prophylactic treatment | 8 | 6 | 7 | 21
  Prior migraine prophylactic treatment only | 119 | 119 | 120 | 358
  No prior / current migraine prophylactic treatment | 192 | 192 | 192 | 576
Monthly Migraine Days [Mean (Standard Deviation); unit: migraine days/month] — A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase. Population: Participants with non-missing values
  migraine days/month
    number analyzed (Participants) | 318 | 316 | 319 | 953
    (all) | 8.23 (2.51) | 8.29 (2.47) | 8.34 (2.48) | 8.29 (2.48)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days to the Last 3 Months of the Double-blind Treatment Period
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine with or without aura.
  The change from baseline in monthly migraine days was calculated as the average number of migraine days per month during the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment phase - the number of migraine days during the 4-week baseline phase.
Time Frame: 4-week baseline phase and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set which includes participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in monthly migraine days in the double-blind treatment phase.
Measure: Least Squares Mean (Standard Error); unit: migraine days / month
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM
Number analyzed (Participants) | 316 | 312 | 318
migraine days / month | -1.83 (0.18) | -3.23 (0.18) | -3.67 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; The primary endpoint was analyzed using a generalized linear mixed model which includes treatment, visit, treatment by visit interaction, stratification factors (region and prior/current treatment with migraine prophylactic medication), and baseline value as covariates; Test type: Superiority — The primary endpoint was tested independently for each erenumab dose at an alpha level of 0.04 for 70 mg and of 0.01 for 140 mg to maintain the type 1 error rate at an alpha level of 0.05; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -1.40, 95% CI 2-sided [-1.88 to -0.92]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 140 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -1.85, 95% CI 2-sided [-2.33 to -1.37]

2. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Monthly Migraine Days in the Last 3 Months of the Double-blind Treatment Phase
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura.
  At least a 50% reduction from baseline in monthly migraine days was determined if the change in monthly migraine days from the 4-week baseline phase to the last 3 months (mean of months 4, 5 and 6) of the 24-week double-blind treatment phase * 100 / baseline monthly migraine days was less than or equal to -50%.
Time Frame: 4-week baseline phase and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set which includes participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in monthly migraine days in the double-blind treatment phase. Participants with missing data at months 4, 5, and 6 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM
Number analyzed (Participants) | 316 | 312 | 318
percentage of participants | 26.6 | 43.3 | 50.0
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; Analyzed using a Cochran-Mantel-Haenszel test, stratified by the randomization stratification factors (region and prior/current treatment with migraine prophylactic medication); Test type: Superiority — If the primary endpoint was statistically significant for the erenumab 70 mg group, using a gate-keeping strategy, the first two (first tier) secondary endpoints were tested using the Hochberg method at an alpha level of 0.04; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.52 to 2.98]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 140 mg QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — If the primary endpoint was statistically significant for the erenumab 140 mg group, using a gate-keeping strategy, the first two (first tier) secondary endpoints were tested using the Hochberg method at an alpha level of 0.01; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.81, 95% CI 2-sided [2.01 to 3.94]

3. Secondary Outcome: Change From Baseline in Monthly Acute Migraine-specific Medication Treatment Days to the Last 3 Months of the Double-blind Treatment Period
Description: Monthly acute migraine-specific medication treatment days is the number of days on which migraine specific medications were used between monthly doses of study drug. Migraine-specific medications includes two categories of medications: triptan-based migraine medications and ergotamine-based migraine medications.
  The change from baseline in monthly acute migraine-specific treatment days was calculated as the average number of migraine-specific treatment days per month during the last 3 months of the 24-week double-blind treatment phase - the number of migraine-specific treatment days during the 4-week baseline phase.
Time Frame: 4-week baseline phase and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set which includes participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in monthly acute migraine-specific treatment days in the double-blind treatment phase.
Measure: Least Squares Mean (Standard Error); unit: Acute migraine-specific med days/mo
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM
Number analyzed (Participants) | 316 | 312 | 318
Acute migraine-specific med days/mo | -0.20 (0.11) | -1.13 (0.11) | -1.61 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; Analyzed using a generalized linear mixed model which includes treatment, visit, treatment by visit interaction, stratification factors (region and prior/current treatment with migraine prophylactic medication), and baseline value as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -0.94, 95% CI 2-sided [-1.23 to -0.64]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 140 mg QM; Analyzed using a generalized linear mixed model which includes treatment, visit, treatment by visit interaction, (stratification factors region and prior/current treatment with migraine prophylactic medication), and baseline value as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -1.42, 95% CI 2-sided [-1.71 to -1.12]

4. Secondary Outcome: Change From Baseline in Mean Monthly Average Physical Impairment Domain Score Measured by MPFID in the Last 3 Months of the Double-blind Treatment Phase
Description: The Migraine Physical Function Impact Diary (MPFID) is a self-administered 13-item instrument measuring physical functioning. It has two domains, Impact on Everyday Activities (7 items) and Physical Impairment (5 items), and one stand-alone global question. Participants completed the MPFID daily in an electronic diary based on the past 24 hours. Participants responded to each item on a 5-point scale, with difficulty items ranging from "Without any difficulty" (1) to "Unable to do" (5) and frequency items ranging from "None of the time" (1) to "All of the time" (5). For each domain, the scores were calculated as the sum of the responses and rescaled to 0 - 100, with higher scores representing greater impact of migraine.
  Change from baseline was calculated as (mean monthly average physical impairment scores as measured by the MPFID over the last 3 months of the double-blind treatment period) - (baseline monthly average physical impairment scores as measured by the MPFID).
Time Frame: 4-week baseline phase and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set including participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in MPFID average physical impairment domain score in the double-blind treatment phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM
Number analyzed (Participants) | 316 | 312 | 318
units on a scale | -2.38 (0.40) | -4.24 (0.40) | -4.81 (0.40)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg QM; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — If the first tier secondary endpoints were statistically significant for both erenumab doses the erenumab 140 mg group for the 2 remaining MPFID secondary endpoints was tested using the Hochberg method at a level of 0.05; If only the erenumab 70 mg group or 140 mg group showed statistical significance for the first tier secondary endpoints then the erenumab 140 group for the 2 remaining MPFID secondary endpoints was tested for significance at a level of either 0.04 or 0.01 respectively; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -2.43, 95% CI 2-sided [-3.51 to -1.35]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 70 mg QM; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — If the erenumab 140 mg group for both remaining MPFID secondary endpoints were statistically significant, then the erenumab 70 mg group for the two remaining MPFID secondary endpoints was tested for significance using the Hochberg method with the same alpha level carried over from 140 mg group; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -1.86, 95% CI 2-sided [-2.95 to -0.77]

5. Secondary Outcome: Change From Baseline in Mean Monthly Average Impact on Everyday Activities Score Measured by MPFID in the Last 3 Months of the Double-blind Treatment Phase
Description: The Migraine Physical Function Impact Diary (MPFID) is a self-administered 13-item instrument measuring physical functioning. It has two domains, Impact on Everyday Activities (7 items) and Physical Impairment (5 items), and one stand-alone global question. Participants completed the MPFID daily in an electronic diary based on the past 24 hours. Participants responded to each item on a 5-point scale, with difficulty items ranging from "Without any difficulty" (1) to "Unable to do" (5) and frequency items ranging from "None of the time" (1) to "All of the time" (5). For each domain, the scores were calculated as the sum of the responses and rescaled to 0 - 100, with higher scores representing greater impact of migraine.
  Change from baseline was calculated as (mean monthly impact on everyday activities scores as measured by the MPFID over the last 3 months of the double-blind treatment period) - (baseline monthly impact on everyday activities scores as measured by the MPFID).
Time Frame: 4-week baseline phase and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment phase
Population: The analysis was conducted in the efficacy analysis set including participants who received at least 1 dose of study drug and had at least 1 change from baseline measurement in MPFID average impact on everyday activities domain score in the double-blind treatment phase.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Erenumab 70 mg QM | Erenumab 140 mg QM
Number analyzed (Participants) | 316 | 312 | 318
units on a scale | -3.30 (0.39) | -5.52 (0.39) | -5.86 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 140 mg QM; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -2.57, 95% CI 2-sided [-3.62 to -1.51]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 70 mg QM; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -2.22, 95% CI 2-sided [-3.28 to -1.16]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 16 weeks after the last dose. The double-blind treatment phase was 24 weeks and the open-label treatment phase was 28 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Double-blind Treatment Phase: Placebo: Participants received placebo once a month (QM) by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase.
- Double-blind Treatment Phase: Erenumab 70 mg: Participants received erenumab 70 mg QM by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase.
- Double-blind Treatment Phase: Erenumab 140 mg: Participants received erenumab 140 mg QM by subcutaneous injection on day 1 and weeks 4, 8, 12, 16, and 20 in the 24-week double-blind treatment phase.
- Active Treatment Phase: Erenumab 70 mg: Participants received erenumab 70 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
- Active Treatment Phase: Erenumab 140 mg: Participants received erenumab 140 mg subcutaneously at weeks 24, 28, 32, 36, 40, 44, and 48 in the active treatment phase.
Arm/Group | Double-blind Treatment Phase: Placebo | Double-blind Treatment Phase: Erenumab 70 mg | Double-blind Treatment Phase: Erenumab 140 mg | Active Treatment Phase: Erenumab 70 mg | Active Treatment Phase: Erenumab 140 mg
Serious Adverse Events (participants affected / at risk) | 7/319 | 8/314 | 8/319 | 14/421 | 14/424
Other Adverse Events (participants affected / at risk) | 53/319 | 53/314 | 54/319 | 83/421 | 63/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Phase: Placebo (N=319) | Double-blind Treatment Phase: Erenumab 70 mg (N=314) | Double-blind Treatment Phase: Erenumab 140 mg (N=319) | Active Treatment Phase: Erenumab 70 mg (N=421) | Active Treatment Phase: Erenumab 140 mg (N=424)
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Arrhythmogenic right ventricular dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Idiopathic orbital inflammation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Prolactin-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Cerebral venous thrombosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Phase: Placebo (N=319) | Double-blind Treatment Phase: Erenumab 70 mg (N=314) | Double-blind Treatment Phase: Erenumab 140 mg (N=319) | Active Treatment Phase: Erenumab 70 mg (N=421) | Active Treatment Phase: Erenumab 140 mg (N=424)
Upper respiratory tract infection (Infections and infestations) | 19 | 21 | 15 | 25 | 19
Viral upper respiratory tract infection (Infections and infestations) | 34 | 32 | 39 | 58 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.